CLINICAL TRIAL: NCT01426425
Title: ICY-AVNRT (Intracardiac CrYoablation for AtrioVentricular Nodal Reentrant Tachycardia)
Brief Title: Intracardiac CrYoablation for AtrioVentricular Nodal Reentrant Tachycardia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICY-AVNRT
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: AtrioVentricular Nodal Reentrant Tachycardia; Supraventricular Tachycardia; Heart Disease
Keywords: Cardiac cryoablation; AVNRT; heart disease; tachycardia; AtrioVentricular Nodal Reentrant Tachycardia; Supraventricular tachycardia; SVT
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry; Tachycardia, Supraventricular; Heart Diseases; Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryoablation (Experimental): Subjects diagnosed with atrioventricular nodal reentrant tachycardia and treated by cryoablation with Freezor Xtra.
  Interventions: Device: Freezor Xtra Cryoablation Catheter

INTERVENTIONS:
Device: Freezor Xtra Cryoablation Catheter — Freezor® Xtra Cardiac CryoAblation applied for cryoablation of the conducting tissues of the heart in the treatment of patients with atrioventricular nodal reentrant tachycardia using an endocardial approach.

SUMMARY:
ICY-AVNRT (Intracardiac CrYoablation for AtrioVentricular Nodal Reentrant Tachycardia) is a prospective multi-center, nonrandomized, single arm, controlled, unblinded, investigational clinical study. The purpose of this clinical study is to demonstrate the safety and effectiveness of the Freezor® Xtra Cardiac CryoAblation Catheter for the cryoablation of the conducting tissues of the heart in the treatment of patients with atrioventricular nodal reentrant tachycardia (AVNRT) using an endocardial approach.

ELIGIBILITY:
Pre-Electrophysiology Study Inclusion Criteria:

* Supraventricular tachycardia (SVT) compatible with atrioventricular nodal reentrant tachycardia (AVNRT), documented by ECG, TTM, Holter or event monitor

Pre-Electrophysiology Study Exclusion Criteria:

* History of sustained (≥30 seconds) of ventricular tachycardia
* Atrial tachycardia or other arrhythmia that could be confused with AVNRT
* Reversible cause of SVT
* History of previous AVNRT ablation
* Therapy with amiodarone within last 90 days
* Unstable angina/myocardial infarction/open heart surgery in past 60 days
* New York Heart Association (NYHA) Classification III or IV currently or within the past 90 days
* Implantable cardiac rhythm device
* Atrioventricular block (first degree (PR interval ≥ 220ms), second degree, or third degree) or left bundle branch block
* Stroke or transient ischemic attack within the past 180 days
* Life expectancy less than 12 months
* Female known to be pregnant
* Unable/unwilling to give informed consent
* Unable/unwilling to comply with follow-up visits and study requirements
* Less than 18 years of age
* Active systemic infection
* Cryoglobulinemia
* Other conditions where the manipulation of the catheter would be unsafe (for example, intracardiac mural thrombus)
* Participating in a concurrent clinical study that may confound the results of this study

Post-Electrophysiology Study Inclusion Criteria:

* Subject must have one electrophysiology study documented inducible sustained (greater than or equal to 15 seconds) supraventricular tachycardia that is classified as AVNRT.

Post-Electrophysiology Study Exclusion Criteria:

* Presence of a second inducible arrhythmia that could be confused with AVNRT during follow-up or will likely result in ablation within the next 6 months
* Presence of inducible sustained ventricular tachycardia or fibrillation
* Presence of an accessory pathway
* Presence of abnormal conduction or refractoriness parameters of the atrioventricular conduction system.
* Indication for a pacemaker, defibrillator or cardiac resynchronization therapy (CRT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2012-05; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wells, M.D., Principal Investigator — Baylor Univ Medical Ctr Dallas, TX.
Locations (34):
- United States (26):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Pacific Heart Institute, Santa Monica, California
  - Stanford Hospital and Clinics, Stanford, California
  - Baptist Hospital of Miami, Miami, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Park Nicollet Institute, Saint Louis Park, Minnesota
  - Healtheast St. Joseph's Hospital, Saint Paul, Minnesota
  - Southside Hospital, Bay Shore, New York
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Miami Valley Cardiologists, Dayton, Ohio
  - Sacred Heart Medical Center, Springfield, Oregon
  - Capital Cardiovascular Associates, Camp Hill, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Wellmont Cardiovascular Heart Institute, Kingsport, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - St. Luke's Episcopal, Houston, Texas
  - Baylor Research Institute, Plano, Texas
  - Virginia Heart, Falls Church, Virginia
- Canada (8):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Victoria Cardiac Arrhythmia Trials, Inc., Victoria, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hopital du Sacre Coeur de Montreal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
  - Prairie CardioVascular Research Network, Regina, Saskatchewan

REFERENCES:
- [Derived] Wells P, Dubuc M, Klein GJ, Dan D, Roux JF, Lockwood E, Sturmer M, Dunbar D, Novak P, Rao A, Peterson BJ, Kueffer F, Ellenbogen KA; ICY-AVNRT Investigators. Intracardiac ablation for atrioventricular nodal reentry tachycardia using a 6 mm distal electrode cryoablation catheter: Prospective, multicenter, North American study (ICY-AVNRT STUDY). J Cardiovasc Electrophysiol. 2018 Jan;29(1):167-176. doi: 10.1111/jce.13367. Epub 2017 Nov 10. PMID 29044787

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-seven (37) centers (8 in Canada, 29 in the US) confirmed participation in the study, with enrollments having occurred at 34 of those centers. First study enrollment occurred on 14-MAY-2012 and the last enrollment occurred on 25-FEB-2015.
Groups:
- All Participants: All subjects enrolled into the study.
Period: Overall Study
Arm/Group | All Participants
Started | 572
EP Study | 550 (EP study used to assess inclusion and exclusion criteria.)
Intent to Treat | 399 (Met all inclusion and no exclusion criteria.)
Completed | 397 (The pre-specified modified intent-to-treat analysis set was used for the primary objectives.)
Not Completed | 175
Not completed — Exited prior to EP study | 22
Not completed — Inclusion/exclusion criteria not met | 151
Not completed — Met inclusion/exclusion, not treated | 2

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) set consists of subjects who signed the ICY-AVNRT consent form and met all Pre-EP and Post-EP study inclusion and no exclusion criteria who had a Freezor Xtra Cardiac Cryoablation Catheter inserted into the vasculature for the purpose of the ICY-AVNRT study.
Groups:
- mITT Set: The modified intent-to-treat (mITT) set.
Arm/Group | mITT Set
Number analyzed (Participants) | 397
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 279
  Male | 118
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Subject/physician chose not to provide information | 10
  Not reportable per local laws or regulations | 0
  American Indian or Alaska Native | 1
  Asian | 10
  Black or African American | 16
  Hispanic or Latino | 4
  Native Hawaiian or Pacific Islander | 0
  White or Caucasian | 353
  Two or more races | 1
  Other race | 2

OUTCOME MEASURES:

1. Primary Outcome: Chronic Effectiveness (Through 6 Months) of the Freezor Xtra Catheter for the Treatment of AVNRT Using an Endocardial Approach.
Description: Subjects must have met both of the following acute and chronic conditions to be considered a chronic effectiveness (treatment) success:
  * Acute Success: The inability to induce more than one echo beat by the same pacing maneuvers that induced AVNRT before cryoablation (with drug provocation if required for induction before cryoablation) at the conclusion of the study cryoablation procedure assessment.
  * Chronic Success: Lack of documented recurrence of clinical AVNRT during the 6-month follow-up period after the study cryoablation procedure.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | mITT Set
Number analyzed (Participants) | 397
Participants
  Chronic effectiveness success | 368
  Chronic effectiveness failure | 29
Statistical Analysis 1: Comparison: mITT Set; The following hypothesis was tested at a one-sided 0.025 significance level. Ho: PE ≤ 0.83 Ha: PE > 0.83 Where PE is the probability of a subject achieving chronic effectiveness success at the 6-month follow-up and 0.83 (83%) is the pre-specified performance goal; Test type: Superiority or Other; p < 0.0001, Kaplan-Meier log-log 95% CI; Chronic effectiveness prob at 6 months = 0.926, 95% CI 2-sided [0.895 to 0.948] — The chronic effectiveness success probability at 6 months was estimated using the Kaplan-Meier method. The standard error was approximated using Greenwood's formula. A two-sided 95% log-log confidence interval for the probability was constructed

2. Primary Outcome: Chronic Safety (Through 6 Months) of the Freezor Xtra Catheter When Used for the Treatment of AVNRT Using an Endocardial Approach.
Description: Subjects who had at least one safety event during or after their cryoablation procedure or through 6 months of follow-up are considered a primary (chronic) safety failure. A safety event is defined as the occurrence of any adverse event that is adjudicated by the AE Adjudication Committee as being serious and study ablation procedure-related and/or Freezor Xtra Catheter related that: 1) Resulted in death, 2) Resulted in a life-threatening illness or injury, 3) Resulted in permanent impairment of a body function or permanent damage to a body structure, 4) Necessitated significant intervention, such as major surgery or even intravenous medical therapy (e.g., vasopressors), to prevent permanent impairment of a body function or permanent damage to a body structure, or 5) Required in-patient hospitalization or a prolongation of an existing hospital stay.
Time Frame: 6 Months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | mITT Set
Number analyzed (Participants) | 397
Participants
  Chronic safety failure | 4
  Chronic safety success | 393
Statistical Analysis 1: Comparison: mITT Set; The following hypothesis was tested at a one-sided 0.025 significance level. Ho: Ps ≥ 0.07 Ha: Ps < 0.07 Where Ps is the probability of a subject experiencing at least one safety event through 6 months with a 0.07 pre-specified performance goal; Test type: Superiority or Other; p < 0.0001, Kaplan-Meier log-log 95% CI; Safety failure probability at 6 months = 0.01, 95% CI 2-sided [0.004 to 0.027] — The chronic safety failure probability at 6 months was estimated using the Kaplan-Meier method. The standard error was approximated using Greenwood's formula. A two-sided 95% log-log confidence interval for the probability was constructed

3. Secondary Outcome: Chronic Effectiveness (Through 6 Months) of the Freezor Xtra Catheter for the Treatment of AVNRT in Subjects Who Achieved Acute Procedural Success.
Description: If there was no documented evidence of AVNRT recurrence in the post-procedure 6-month follow-up period, the subject is counted as a chronic effectiveness success. The AE Adjudication Committee adjudication of AVNRT recurrence is used to classify subjects for this endpoint.
Time Frame: 6 Months
Population: The 378 mITT subjects who had acute procedural success with cryoablation for the treatment of AVNRT are included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- mITT Subjects With Acute Procedural Success: The modified intent-to-treat (mITT) subjects who had acute procedural success with cryoablation for the treatment of AVNRT.
Arm/Group | mITT Subjects With Acute Procedural Success
Number analyzed (Participants) | 378
Participants
  Chronic effectiveness success | 368
  Chronic effectiveness failure | 10
Statistical Analysis 1: Comparison: mITT Subjects With Acute Procedural Success; The following hypothesis was tested at a one-sided 0.025 significance level. Ho: PE ≤ 0.80 Ha: PE > 0.80 Where PE is the probability of a subject achieving chronic effectiveness success at 6-month follow-up, and 0.80 is the pre-specified performance goal. As pre-defined in the study protocol, this hypothesis is tested if the primary effectiveness objective null hypothesis (Ho) is rejected; Test type: Superiority or Other; p < 0.0001, Kaplan-Meier log-log 95% CI; Chronic effectiveness prob at 6 months = 0.973, 95% CI 2-sided [0.950 to 0.985] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from the time of their enrollment through the visit cut-off date for the primary endpoint analyses (September 18, 2015).
Description: Adverse event information was provided by the investigators. All adverse events were reviewed and adjudicated by an independent (i.e., non-Medtronic) Adverse Events Adjudication Committee as serious or non-serious. Adverse events terms were coded using MedDRA 18.0 by Medtronic safety specialists.
Groups:
- mITT Set: Subjects in the modified intent-to-treat (mITT) set.
Arm/Group | mITT Set
Serious Adverse Events (participants affected / at risk) | 30/397
Other Adverse Events (participants affected / at risk) | 197/397
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mITT Set (N=397)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 3 (3)
Device difficult to use (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Retrognathia (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | mITT Set (N=397)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 9 (12)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 6 (6)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Bundle branch block right (Cardiac disorders) | 11 (11)
Cardiac flutter (Cardiac disorders) | 1 (1)
Junctional ectopic tachycardia (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 43 (55)
Sinus tachycardia (Cardiac disorders) | 7 (7)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 22 (27)
Tachycardia (Cardiac disorders) | 7 (7)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1)
Laryngocele (Congenital, familial and genetic disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 4 (4)
Hypothyroidism (Endocrine disorders) | 2 (2)
Cataract (Eye disorders) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Crohn's disease (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 3 (3)
Chest discomfort (General disorders) | 6 (8)
Chest pain (General disorders) | 18 (19)
Fatigue (General disorders) | 4 (4)
Gait disturbance (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4)
Oedema peripheral (General disorders) | 3 (3)
Pain (General disorders) | 2 (2)
Polyp (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 4 (8)
Bacterial vaginosis (Infections and infestations) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 9 (9)
Cellulitis (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3)
Pharyngitis (Infections and infestations) | 5 (5)
Pharyngitis streptococcal (Infections and infestations) | 3 (4)
Pneumonia (Infections and infestations) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 5 (6)
Skin candida (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (9)
Urinary tract infection (Infections and infestations) | 6 (9)
Vaginal infection (Infections and infestations) | 1 (2)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Animal scratch (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 5 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood iron decreased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 2 (2)
Heart rate increased (Investigations) | 3 (3)
Heart rate irregular (Investigations) | 1 (1)
Hepatitis B antibody positive (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Sinus rhythm (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Zinc deficiency (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint lock (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 3 (3)
Dizziness (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 8 (8)
Loss of consciousness (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 3 (6)
Paraesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 6 (6)
Bipolar disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Madarosis (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (3)
Hypertension (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, the contract allows the principal investigator to publish their data per the publication strategy/Clinical Investigational Plan following Medtronic's review for (a) disclosure of confidential information ("CI"), (b) technical correctness and (c) selection and order of publications by the publications committee. Any such CI and/or item identified as not technically correct is deleted prior to publication/presentation. Medtronic may not otherwise interfere with the publication.